CLINICAL TRIAL: NCT04120285
Title: Remote Cognitive Behavior Therapy for Major Depression (RTD) in Primary Care
Brief Title: Appalachian Mind Health Initiative
Acronym: AMHI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Robert Bossarte, Professor, Department of Psychiatry and Behavioral Neuroscience, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS-2017C3-9252
Record Dates: First submitted 2019-05-31; First posted 2019-10-09 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression; eCBT
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: There are three treatment arms: 1) treatment as usual 2) treatment as usual with unguided eCBT and 3) treatment as usual with guided eCBT
Masking Description: Participant recruiters will be blinded to the participant's intended treatment arm.
  Survey data collectors will be blinded to each participant's treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Primary Care Treatment (No Intervention): The participant will receive treatment as usual as prescribed by the primary care physician for MDD.
- Primary care treatment with eCBT (Active Comparator): The participant will receive treatment as usual as prescribed by the primary care physician with the addition of eCBT for MDD.
  Interventions: Behavioral: remote internet-based cognitive behavior therapy (eCBT)
- Primary care treatment with guided eCBT (Active Comparator): The participant will receive treatment as usual as prescribed by the primary care physician with the addition of guided eCBT for MDD.
  Interventions: Behavioral: remote internet-based cognitive behavior therapy (eCBT)

INTERVENTIONS:
Behavioral: remote internet-based cognitive behavior therapy (eCBT) — Provide access to online psychotherapy program to participants in rural WV areas at no expense to them.
  Arms: Primary care treatment with eCBT; Primary care treatment with guided eCBT

SUMMARY:
We propose to carry out a treatment experiment in which we evaluate the extent to which randomizing primary care clinicians have access to remote internet-based Cognitive Behavior Therapy (eCBT) in rural West Virginia (WV) and Kentucky (KY) will help improve treatment of patients with Major Depressive Disorder (MDD). WV and KY are two of the most rural states in America and mental health treatment resources are low; especially in rural parts of the state.

DETAILED DESCRIPTION:
The investigators propose a pragmatic trial of the comparative effectiveness of two levels of remote internet-based cognitive behavior therapy (eCBT) to treat major depressive disorder (MDD) with and without comorbidities. The investigators intend to recruit 3,360 patients receiving primary care MDD treatment throughout West Virginia (WV) and Kentucky (KY). The investigators two main aims will be to use experimental methods to evaluate the aggregate effects of these interventions on patient-centered outcomes and to investigate predictors of heterogeneity of treatment effects. MDD treatment in WV & KY is far from optimal, with rural patients especially underserved. WV is the 2nd most rural state in the US, has the 2nd lowest per capita income and has the highest proportion of residents covered by Medicaid. Need for services is high, as indicated by WV having the highest suicide rate of any state east of the Mississippi River and the highest opioid death rate in the country. Yet WV ranks only 42nd in overall mental health care. The vast majority of MDD treatment in rural areas is in primary care and consists largely of antidepressant medication (ADM). Electronic medical records (EMRs) show that 88% of primary care MDD patients in WV's FQHCs are treated exclusively with ADM and that the other 12% are treated with ADM plus psychotherapy. The limited number of patients who can access psychotherapy usually must go on a waiting list (often 3+ months) and travel long distances for treatment once available. Access to telephone or videoconference psychotherapy is limited. Yet 75% of depressed primary care patients express a desire for psychotherapy either alone (40%) or in combination with ADM (35%).

This mismatch between treatment availability and preference is important because MDD remission increases substantially when patients are treated with their preferred type. There is thus good reason to believe that providing access to eCBT will improve MDD treatment outcomes in our trial. Indeed, prior controlled trials show that both types of eCBT the investigators will randomize yield significantly better outcomes than waiting list controls. Controlled trials also show that guided eCBT yields equivalent outcomes to telephone and face-to-face CBT, but at much lower cost. Other controlled trials show that combined CBT-ADM yield significantly better outcomes than either CBT-alone or ADM-alone, although these comparisons have been made only for face-to-face CBT. These results provide good reason to believe that offering eCBT in rural FQHCs throughout WV and KY could improve MDD outcomes. Existing research on eCBT in rural areas, while promising, has been limited, making the research the investigators propose important to provide actionable information for patients and other stakeholders. Results intend to inform decisions about whether to offer/use eCBT, with what level of guidance, and for whom.

Unguided eCBT is web-based CBT completed with computerized feedback but no clinician involvement after an initial orientation meeting. Guided eCBT is web-based CBT completed with a remote eCoach who communicates with the patient via email, text, and telephone. eCoaches also provide elements of remote collaborative care case management, such as encouraging ADM adherence, monitoring ADM side effects and treatment response, coordinating with the primary care physician (PCP), and facilitating specialty referral. Collaborative care is known to be highly effective in promoting MDD symptomatic remission. In addition, a study in Arkansas FQHCs found that remote collaborative care case management out-performed on-site case management in rural clinics too small to justify having a dedicated mental health case manager on staff. However, remote collaborative care case management often involves delivering telephone CBT. A major constraint on expanding the collaborative care model for primary care MDD treatment, which has been used in urban but not rural WV clinics, is lack of case managers who can deliver telephone CBT. Thus, expanding eCBT in rural WV would allow offering a strongly evidence-based form of patients' preferred treatment (psychotherapy) and a form of a well-validated rural MDD care model (collaborative care case management with guided eCBT) that cannot be offered currently because of limited clinical resources.

Given its documented efficacy and rapid spread, the investigators expect eCBT to become widely available in rural WV as a result of our trial. But two real-life decisional dilemmas will arise in that context. Primary care clinicians will be faced with the decision about when to recommend eCBT and at what level of intensity. Patients will be faced with the decision of whether to accept guided or unguided eCBT as part of their treatment plan. These are non-trivial decisions, as eCBT incurs a time cost, and guided eCBT incurs a financial cost and requires interactions with a supporter for patients who desire independence and privacy. Further, eCBT has the potential to harm, as when lack of engagement leads the patient to drop out of all treatment, including ADM, whereas that patient would have remitted with ADM. Our heterogeneity of treatment effects (HTE) analyses will examine which patients profit from guided eCBT, which do equally well or better with unguided than guided eCBT, and which do as well or better with ADM in the absence of eCBT. A good deal of research has been carried out on eCBT HTE, although not in conjunction with ADM. This research suggests that the value of eCBT for MDD varies considerably depending on diverse patient characteristics the investigators plan to study. As with the comparative effectiveness evidence for eCBT vs other MDD therapies, though, research on MDD HTE up to now has focused on narrowly-defined symptom outcomes. In addition, although more than two dozen consistently significant baseline patient-reported predictors of MDD HTE have been documented, no single study ever considered more than a handful of these predictors. In addition, past MDD HTE studies have been underpowered. Our analysis will be based on a sample of 3,360 patients powered to detect HTE in the entire sample. Our patient and provider partners have indicated that evidence about the prescriptive predictors of these differences will be of great value in their treatment selection decisions. The causal model underlying the design is drawn from previous studies reviewed here: that MDD remission of primary care patients can be increased by adding eCBT to treatment-as-usual (TAU) via mechanisms that include influencing cognitions and behaviors to promote psychological recovery and encouraging increased ADM compliance. This model underlies all aspects of our design (selection of population, interventions, measures, analytic methods, procedures for handling confounding, time frame).

ELIGIBILITY:
Inclusion criteria:

1. seeking MDD treatment for the first time in the past 6 months (i.e., the beginning of a first or new course of treatment),
2. appropriate for outpatient treatment,
3. literate in English,
4. has access to a smart phone, home computer or willing to travel to access a computer
5. without hearing or vision or cognitive impairment that would interfere with research data collection
6. without history of either bipolar disorder or non-affective psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3360 (Estimated)
Dates: Start 2021-01-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
RDQ-7 | 16-Week Follow-up
  Investigators will assess all study patients remission from depression with the Remission from Depression Questionnaire (RDQ-7) via self-report assessments at 16 week follow-up. Investigators will monitor patients at 26, 39, and 52 weeks to evaluate the long-term maintenance of remission (or recurrence). The RDQ-7 is a measure with 41 items. Items are reported on a 3-point rating scale (0=not at all or rarely true; 1 = sometimes; 2 = often or almost always true). The total scale score ranges from 0-82. Participants with a total score below or equal to 27 are considered in remission. Higher total scores reflect greater pathology.

SECONDARY OUTCOMES:
PROMIS Short Form v1.0 - Severity of Substance Use (past 30 days) | 16 week Follow-up
  The investigators will assess all study participants severity of substance use using the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Severity of Substance Use (past 30 days) at 16 week follow-up. Investigators will monitor participants at 26, 39, and 52 weeks to evaluate the long-term durability of our intervention. The PROMIS) Short Form v1.0 - Severity of Substance Use (past 30 days) is a measure with 7 items. Items are reported with five response options ranging in value from one to five. To calculate the total scale score, items are summed resulting in a range from 1-35. Higher total scores reflect that a participant uses a substance with greater severity.
Compliance with Antidepressant Medication Treatment | 16 week Follow-up
  The investigators will assess all study participants adherence to antidepressant medication (if applicable) using electronic medical record data at 16 week follow-up. Investigators will monitor participants at 26, 39, and 52 weeks to evaluate the long-term durability of our intervention. Electronic medical record data will be examined for antidepressant medication prescriptions and prescription refills or changes.
SDM-Q-9 | 52 week Follow-up
  The investigators will assess all study participants involvement with shared decision-making regarding depression treatment provided by their primary care physician using the Shared Decision Making Questionnaire (SDM-Q-9) at 52 week follow-up. The SDM-Q-9 is a nine item measure. Items are reported with six response options ranging from 0, "completely disagree", to 5, "completely agree". To calculate the total scale score, items are summed resulting in a range from 0-45. Higher scores reflect a participant's participation in shared decision making regarding their treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bossarte, PhD, Principal Investigator — University of South Florida; Ronald Kessler, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (7):
- United States (7):
  - University of Lousiville Health, Louisville, Kentucky
  - Upper Kanawha Clinic, Cedar Grove, West Virginia
  - Minnie Hamilton Health Systems, Glenville, West Virginia
  - Minnie Hamilton Health Systems, Grantsville, West Virginia
  - Harpers Ferry Family Medicine, Harpers Ferry, West Virginia
  - WVU Medicine, Morgantown, West Virginia
  - Wayne Medical Clinic, Wayne, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bossarte RM, Kessler RC, Nierenberg AA, Chattopadhyay A, Cuijpers P, Enrique A, Foxworth PM, Gildea SM, Belnap BH, Haut MW, Law KB, Lewis WD, Liu H, Luedtke AR, Pigeon WR, Rhodes LA, Richards D, Rollman BL, Sampson NA, Stokes CM, Torous J, Webb TD, Zubizarreta JR. The Appalachia Mind Health Initiative (AMHI): a pragmatic randomized clinical trial of adjunctive internet-based cognitive behavior therapy for treating major depressive disorder among primary care patients. Trials. 2022 Jun 20;23(1):520. doi: 10.1186/s13063-022-06438-y. PMID 35725644